CLINICAL TRIAL: NCT01266655
Title: Baclofen for the Treatment of Alcohol Dependence - BACLAD
Brief Title: Baclofen for the Treatment of Alcohol Dependence
Acronym: BACLAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. A. Heinz, M.D., Department of Psychiatry, Charité Campus Mitte, Charité - Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BACLAD
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen (Experimental)
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Baclofen will be administered orally for a maximum of 20 consecutive weeks. For the first 3 days, patients will receive baclofen in a dose of 5 milligrams t.i.d.; subsequently, the daily dose of baclofen will be increased to a maximum of 90 milligrams t.i.d. within 4 weeks. In case of intolerance, dosage can be decreased to a minimum of 10 mg t.i.d.. Patients will receive maximum tolerated dosage of baclofen for 12 weeks. Medication will then gradually be tapered over a maximum of 4 weeks.
  Arms: Baclofen
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
There is first evidence from preclinical and clinical studies for the efficacy of the selective GABA-B receptor agonist baclofen in the treatment of alcohol dependence. The aim of this trial is to evaluate the efficacy and safety of individually titrated high-dose baclofen for relapse prevention in alcohol-dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol dependence according to ICD-10 (International Classification of Mental and Behavioural Disorders, 10th revision) and DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th revision) criteria
* An alcohol intake of at least two heavy drinking days per week on average (men ≥ 5 drinks per day; women ≥ 4 drinks per day) and an average overall consumption of 21 drinks per week or more for men and 14 drinks per week or more for women during the 4 weeks before detoxification (one standard drink is equal to 12 g absolute alcohol)
* Last alcohol consumption within 7-21 days before randomisation
* Sufficient German language capabilities

Exclusion Criteria:

* Pregnancy and/or currently breastfeeding
* Clinical significant medical conditions or observed abnormalities
* Psychiatric illness undergoing treatment with psychoactive drugs
* Epilepsy or epileptiform convulsions
* Addiction to drugs other than nicotine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Total abstinence from alcohol and cumulative abstinence duration | 13-16 weeks (depending on the individually tolerated baclofen dose)

SECONDARY OUTCOMES:
Number of adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Heinz, Prof., M.D., Principal Investigator — Department of Psychiatry, Charité Campus Mitte, Charité - Universitätsmedizin Berlin, Germany
Locations (1):
- Department of Psychiatry, Charité Campus Mitte, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Beck A, Pelz P, Lorenz RC, Charlet K, Geisel O, Heinz A, Wustenberg T, Muller CA. Effects of high-dose baclofen on cue reactivity in alcohol dependence: A randomized, placebo-controlled pharmaco-fMRI study. Eur Neuropsychopharmacol. 2018 Nov;28(11):1206-1216. doi: 10.1016/j.euroneuro.2018.08.507. Epub 2018 Sep 11. PMID 30217552